CLINICAL TRIAL: NCT05343078
Title: Pharmacokinetics and Dialyzability of Dapagliflozin in Dialysis Patients: on Behalf of the DARE-ESKD Trial
Brief Title: Pharmacokinetics and Dialyzability of Dapagliflozin in Dialysis Patients
Acronym: DARE-ESKD 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, Chairman of the Clinical Research Center, University of Campinas, Brazil
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 50393421.4.0000.5404
Record Dates: First submitted 2022-04-07; First posted 2022-04-25 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: End-stage Renal Disease
Keywords: hemodialysis; dapagliflozin; peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: In the single-dose protocol, hemodialysis participants will take the experimental drug immediately prior to the dialysis session. In the multiple-dose protocol, volunteers will take the drug daily in the morning for one week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dapagliflozin (Experimental): Dapagliflozin 10mg P.O.
  Interventions: Drug: Dapagliflozin 10Mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — Participants will take a single-dose Dapagliflozin 10mg P.O. prior to the hemodialysis session for the single-dose pharmacokinetics protocol. In the multiple-dose protocol, Dapagliflozin 10mg P.O. will be taken daily in the morning for one week.

SUMMARY:
Sodium-glucose co-transporter 2 inhibitors (Sglt2i) attenuate the incidence of cardiovascular events in individuals with preserved or mildly reduced kidney function. Whether this benefit is also observed among individuals with end-stage renal disease (ESRD), in whom cardiovascular disease is a leading cause of mortality, remains unexplored. To appraise the influence of dialysis on the pharmacokinetics of Sglt2i is a prerequisite to determining the treatment regimen that best fits this population.

In this study ESRD individuals, aged 18 years and older, on a regular dialysis regimen for a minimum of 3 months at the Nephrology Division of the Clinics Hospital of the University of Campinas (Unicamp) will be enrolled in a pharmacokinetics study.

In the single-dose protocol, hemodialysis participants will take Dapagliflozin 10mg P.O. immediately before the dialysis session, and blood samples will be collected every 30min during dialysis and again 24h and 48h after termination. The dialysate will be continuously sampled in a tank and aliquots collected for further analysis.

In the multiple-dose protocol, both hemodialysis and peritoneal dialysis participants will take Dapagliflozin 10mg P.O. daily in the morning for 7 days. Blood samples will be collected at baseline, and again after 48h and 7 days.

The plasma levels of dapagliflozin and its inactive metabolite, D3OG, will be calculated from blood and dialysate samples using liquid chromatography mass spectrometry.

The primary outcome is the plasma concentration-time curve of dapagliflozin and its inactive metabolite D3OG during a regular hemodialysis session. Secondary outcomes are: (i) the steady-state plasma concentration of Dapa; (ii) the accumulation ratio of Dapa; (iii) the total mass of Dapa and D3OG extracted by the dialysate; (iv) the dialytic clearance of dapagliflozin.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis for 3 months or more prior to enrollment
* 18 years of age or older
* Signed the informed consent form

Exclusion Criteria:

* Liver dysfunction
* Allergy to dapagliflozin
* Currently receiving a Sglt2i

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve of the plasma concentration-time curve of dapagliflozin | From dialysis initiation to 48 hours post- drug administration
  AUC of dapagliflozin (ng.mL / mL)

SECONDARY OUTCOMES:
Area under the curve of the plasma concentration-time curve of D3OG | From dialysis initiation to 48 hours post- drug administration
  AUC of D3OG (ng.mL / mL)
Steady-state plasma concentration of Dapagliflozin | 7 days
  Steady-state plasma concentration (ng/mL)
Steady-state accumulation ratio of Dapagliflozin | 7 days
  Accumulation index
Total mass of dapagliflozin extracted by the dialysis | 7 days
  Dapagliflozin mass (mg)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barreto J, Borges C, Rodrigues TB, Jesus DC, Campos-Staffico AM, Nadruz W, Luiz da Costa J, Bueno de Oliveira R, Sposito AC. Pharmacokinetic Properties of Dapagliflozin in Hemodialysis and Peritoneal Dialysis Patients. Clin J Am Soc Nephrol. 2023 Aug 1;18(8):1051-1058. doi: 10.2215/CJN.0000000000000196. Epub 2023 May 25. PMID 37227937